CLINICAL TRIAL: NCT05891236
Title: A Phase 1, Dose Escalation, Double Blind, Placebo Controlled Clinical Trial With Controlled Human Malaria Infections (CHMI) to Evaluate Safety, Tolerability, Pharmacokinetics, and Protective Efficacy of an Anti-Malaria Human Monoclonal Antibody, MAM01, in Healthy, Malaria-Naive Adults
Brief Title: Safety, Tolerability, Pharmacokinetics and Protective Efficacy of MAM01 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: Gates MRI-MAM01-101
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Malaria
Keywords: Healthy volunteers; MAM01 monoclonal antibody; First-in-Human; Dose-escalation; Single ascending dose; Multiple ascending dose; Recruiting; Malaria vaccine; Mosquito; Gates; Prevention; Phase 1; Nonprofit
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A: Single Ascending Dose (SAD): Dose escalation cohort 1: MAM01 and placebo Intravenous (IV) (Experimental): 2 sentinel participants will be randomized in a 1:1 ratio to receive MAM01 1.5 milligrams per kilogram (mg/kg) IV or placebo. Following at least a 24-hour safety review period, the 6 remaining participants of Cohort 1 will be randomized in a 5:1 ratio to receive MAM01 1.5 mg/kg IV or placebo.
  Interventions: Biological: MAM01 1.5 mg/kg; Biological: Placebo
- Part A: SAD dosing: Dose escalation Cohort 2: MAM01 and placebo SC (Experimental): 7 participants will be randomly assigned in a 6:1 ratio to receive MAM01 5 mg/kg SC or placebo
  Interventions: Biological: MAM01 5 mg/kg; Biological: Placebo
- Part A: SAD dosing: Dose escalation Cohort 3: MAM01 and placebo IV (Experimental): 7 participants will be randomly assigned in a 6:1 ratio to receive MAM01 5 mg/kg IV or placebo.
  Interventions: Biological: Placebo; Biological: MAM01 5 mg/kg
- Part A: SAD dosing: Dose escalation Cohort 4: MAM01 and placebo IV (Experimental): 8 participants will be randomly assigned in a 6:2 ratio to receive MAM01 10 mg/kg IV or placebo.
  Interventions: Biological: Placebo; Biological: MAM01 10 mg/kg
- Part A: SAD dosing: Dose escalation Cohort 5: MAM01 and placebo IV (Experimental): 7 participants will be randomly assigned in a 6:1 ratio to receive MAM01 40 mg/kg IV or placebo
  Interventions: Biological: Placebo; Biological: MAM01 40 mg/kg
- Part A: Multiple Ascending Dose (MAD) (Repeat dosing): MAM01 (Experimental): Participants from Cohort 2 and from Cohort 3 will receive 5 mg/kg MAM01 SC.
  Interventions: Biological: MAM01 5 mg/kg
- Part B: Dose Expansion Cohort 6: Group 1: MAM01 (Experimental): 6 participants will receive a 450 mg SC dose of MAM01. The dose was selected by applying a PK-pharmacodynamic (PD) model from the Part A data to estimate a (data-driven) protection threshold at Controlled Human Malaria Infection (CHMI).
  Interventions: Biological: MAM01 450 mg
- Part B: Dose Expansion Cohort 6: Group 2: MAM01 (Experimental): 8 participants will receive a 600 mg SC dose of MAM01. The dose was selected by applying a PK-PD model from the Part A data to estimate a (data-driven) protection threshold at CHMI
  Interventions: Biological: MAM01 600 mg
- Part B: Dose Expansion Cohort 6: Group 3: MAM01 (Experimental): 8 participants will receive 900 mg SC dose of MAM01. The dose was selected by applying a PK-PD model from the Part A data to estimate a (data-driven) protection threshold at CHMI.
  Interventions: Biological: MAM01 900 mg
- Internal Infectivity Controls (Experimental): 6 participants will be enrolled into a non-randomized group prior to CHMI. These participants will receive no treatment and act as infectivity controls
  Interventions: Other: Control

INTERVENTIONS:
Biological: MAM01 1.5 mg/kg — 1.5 mg/kg MAM01 will be administered via IV route.
  Arms: Part A: Single Ascending Dose (SAD): Dose escalation cohort 1: MAM01 and placebo Intravenous (IV)
Biological: Placebo — Placebo will be administered via IV route.
  Arms: Part A: SAD dosing: Dose escalation Cohort 3: MAM01 and placebo IV; Part A: SAD dosing: Dose escalation Cohort 4: MAM01 and placebo IV; Part A: SAD dosing: Dose escalation Cohort 5: MAM01 and placebo IV; Part A: Single Ascending Dose (SAD): Dose escalation cohort 1: MAM01 and placebo Intravenous (IV)
Biological: MAM01 5 mg/kg — 5 mg/kg MAM01 will be administered via SC route.
  Arms: Part A: Multiple Ascending Dose (MAD) (Repeat dosing): MAM01; Part A: SAD dosing: Dose escalation Cohort 2: MAM01 and placebo SC
Biological: MAM01 10 mg/kg — 10 mg/kg MAM01 will be administered via IV route.
  Arms: Part A: SAD dosing: Dose escalation Cohort 4: MAM01 and placebo IV
Biological: MAM01 40 mg/kg — 40 mg/kg MAM01 will be administered via IV route.
  Arms: Part A: SAD dosing: Dose escalation Cohort 5: MAM01 and placebo IV
Biological: MAM01 450 mg — MAM01 will be administered via SC route.
  Arms: Part B: Dose Expansion Cohort 6: Group 1: MAM01
Biological: Placebo — Placebo will be administered via SC route.
  Arms: Part A: SAD dosing: Dose escalation Cohort 2: MAM01 and placebo SC
Biological: MAM01 5 mg/kg — 5 mg/kg MAM01 will be administered via IV route.
  Arms: Part A: SAD dosing: Dose escalation Cohort 3: MAM01 and placebo IV
Other: Control — No drug or placebo will be administered.
  Arms: Internal Infectivity Controls
Biological: MAM01 600 mg — MAM01 will be administered via SC route.
  Arms: Part B: Dose Expansion Cohort 6: Group 2: MAM01
Biological: MAM01 900 mg — MAM01 will be administered via SC route.
  Arms: Part B: Dose Expansion Cohort 6: Group 3: MAM01

SUMMARY:
This is a First-in-Human (FiH), randomized, two-part, dose-escalation trial of MAM01 monoclonal antibody (mAb) targeting the Plasmodium falciparum (Pf) Circumsporozoite Protein (CSP). This study will evaluate the safety, tolerability, pharmacokinetics (PK), and protective efficacy of MAM01, as well as safety and PK of repeat subcutaneous (SC) dosing. Part A will have a double-blind, placebo-controlled design. Part B will randomize participants to one of three open-label MAM01 dose groups; a separate non-randomized group will be enrolled to include participants who will receive no treatment and act as infectivity controls.

ELIGIBILITY:
Inclusion criteria:

* Participants who are healthy as determined by medical evaluation including medical history, physical examination and laboratory tests
* Body Mass Index (BMI) 18 to 30 kilograms per square meter (kg/m^2) (inclusive) to a maximum of 220 pounds
* Both males and females are eligible to participate as per the following:

  a. Female participants physically capable of pregnancy, have at least one negative pregnancy test during Screening, on the day of enrollment, prior to Investigational product (IP) administration, prior to CHM and at the start of antimalarial treatment, and who agree to use effective contraception to avoid pregnancy from 28 days before enrollment through 10 months after last administration of investigational product are eligible to participate.
* Capable of giving signed Informed Consent which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and the trial protocol, and completion of a test of understanding if he/she may participate in the CHMI procedure
* Reported completion of primary Coronavirus Disease (COVID) vaccine series is documented

Exclusion criteria:

* Acute illness or fever ≥99.5°Fahrenheit (F) (or ≥37.5 degrees Celsius) on day of dosing
* Women who are pregnant or breastfeeding
* Evidence and/or history of clinically significant medical condition(s) as judged by the Investigator, including malignancies, diabetes mellitus, and unstable or uncontrolled hypertension
* A 5-year cardiovascular risk of ≥10% using the Gaziano nomogram
* History of any autoimmune disease or immune deficiency or other impairment to the immune system, including but not limited to Human immunodeficiency virus (HIV), autoimmune conditions or immunosuppressive therapy
* Participation in an interventional clinical trial and/or receipt of any investigational drug within 180 days prior to administration of trial drug on Day 0
* Anticipated use of medications known to cause drug reactions with chloroquine or atovaquone-proguanil (Malarone) such as cimetidine, metoclopramide, antacids, and kaolin

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited local and systemic adverse events (AEs) in the SC cohorts | Through 7 days post-dose
  Local injection site solicited AEs will be assessed after dosing and will also be recorded for 7 days from SC recipients only. Systemic solicited AEs will be assessed in all participants after dosing at Visit 1 and recorded for 7 days.
Number of participants reporting unsolicited AEs (single dose or multiple dose) | Through Day 28
  Unsolicited adverse events will be captured after product administration and the CHMI procedure
Number of participants reporting serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) and adverse events special interest (AESIs) | Through 168 days post-dose
  A SAE is defined as any untoward medical occurrence that, at any dose: Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or is a medically significant / important event or reaction. SUSARs are adverse event that occur in a clinical trial participant, which is assessed by the Sponsor and or study investigator as being unexpected, serious and as having a reasonable possibility of a causal relationship with the study drug. AESIs are adverse events that the Sponsor wants to monitor carefully and which are subject to expedited reporting
Number of re-dosed participants reporting SUSARs, SAEs and AESIs | Through 378 days
Number of participants with safety laboratory assessments by grade (grade 1 and above) | Up to 378 Days
  Blood samples will be collected for the analysis of laboratory parameters including hematology and serum chemistry.

SECONDARY OUTCOMES:
Maximal observed concentration (Cmax) following single and repeat dosing of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via Volumetric Absorptive Microsampling Method (VAMS) or microtainers will be collected from participants in the Pharmacokinetic (PK) Population for measurement of MAM01 Cmax. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Area under the curve (AUC) from Time=0 to the last measurable concentration (AUC0-t) of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 AUC 0-t. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Partial AUC's Time= 0 to the CHMI challenge (AUC0-CHMI) of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 AUC0-CHMI. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Concentration at the time of CHMI (CCHMI) following single and repeat dosing of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 CCHMI. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Blood terminal elimination rate constant (λz) following single and repeat dosing of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 λz. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Terminal half life (t1/2) of MAM01 | Time Frame: Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 t1/2. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
AUC from Time=0 extrapolated to infinity (AUC0-infinity) of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 AUC0-infinity. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Percentage (%) AUC extrapolated (% AUCext) of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 (% AUCext. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Bioavailability of SC formulation following single and repeat dosing of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140, 168, 224 and 280 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 bioavailability. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Part A: Cohorts 2 and 3: Accumulation ratio (AUC0-168) of MAM01 | Pre-dose, Day 0: end of infusion (EOI), 1, 3 and 6 hours, Day 1: 24 hours, Day 2: 48 hours, Days 7, 14, 28, 42, 56, 70, 84, 98, 112, 140 and 168 post-dose
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 AUC0-168. Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Part A: Cohorts 2 and 3: AUC (210-378) of MAM01 | Day 210 and up to Day 378
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 AUC (210-378). Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Part A: Cohorts 2 and 3: Accumulation ratio AUC (210-378) of MAM01 | Day 210 and up to Day 378
  Capillary blood samples via VAMS or microtainers will be collected from participants in the PK Population for measurement of MAM01 Accumulation ratio AUC (210-378). Blood concentrations of MAM01 will be measured using a qualified immunoassay.
Number of participants with presence or absence of Pf infection assessed by quantitative polymerase chain reaction assay (qRT-PCR) after CHMI | Through Day 27 post CHMI
  A sensitive qRT-PCR will be used for the detection of Pf parasites in Efficacy Population.
Time to parasitemia after CHMI in Efficacy Population | Up to Day 378
Part A: Cohorts 1, 4 and 5: Titers of anti-drug antibodies (ADAs) following administration of MAM01 in Immunogenicity Population | Up to Day 280
  Percentage of participants with titers confirmed above the assay cut point will be summarized calculated by treatment group as appropriate.
Part A: Cohorts 2 and 3: Titers of ADAs following administration of MAM01 in Immunogenicity Population | Up to Day 378
Part B: Cohort 6: Titers of Number of participants with ADAs following administration of MAM01 in Immunogenicity Population | Up to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: +1 866 789 5767, Study Director — Gates Medical Research Institute
Locations (1):
- Center for Vaccine Development and Global Health, 685 W. Baltimore Street, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyke KE, Berry AA, Laurens MB, Winkler J, Joshi S, Koudjra AR, Butler L, Billingsley PF, Pascini T, Patil A, Sim BKL, Fitzgerald G, Riegel J, Andrews K, Levi M, Anderson AB, Wells CD, Liu H, Huleatt J, Miller RS. Human monoclonal antibody MAM01 for protection against malaria in adults in the USA: a first-in-human, phase 1, dose-escalation, double-blind, placebo-controlled, adaptive trial. Lancet Infect Dis. 2025 Sep 23:S1473-3099(25)00481-5. doi: 10.1016/S1473-3099(25)00481-5. Online ahead of print. PMID 41005346